CLINICAL TRIAL: NCT02630615
Title: Circulating Tumor Cells (CTC) in Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Shadia Jalal (Other)
Responsible Party: Sponsor-Investigator, Shadia Jalal, Assistant Research Professor, Assistant Professor of Clinical Medicine, Indiana University
Organization: Indiana University (Other)
Other Study IDs: IUSCC-0567; 1512076915 (Other: Indiana University IRB)
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Lung Neoplasms
Keywords: Circulating tumor cells
MeSH Terms: conditions — Lung Neoplasms; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A (one-time blood sample): Blood samples will be collected from eligible patients only once at baseline. These samples will be immediately processed for CTCs and CTC derived xenografts.
  For Cohorts A & B: Patients can participate in both cohorts simultaneously, or only one cohort per patient preference.
  Interventions: Other: Blood draw
- Cohort B (multiple blood samples): Blood samples will be collected from eligible patients at baseline just prior to initiation of therapy. Samples will also be collected on day 1 of every cycle of therapy for 4 cycles (typical cycles are 21 days for chemotherapy, 28 days for targeted therapy and 14 days for immune therapy). At the time of initiation of the treatment break, blood samples will be collected. During the treatment break, patients will be followed every 6-12 weeks with imaging studies, and we will collect blood samples at each visit. At the time of disease progression in the event patient goes on best supportive care, the last blood draw will be at the time of this decision as there will unlikely be any further imaging studies going forward. If a patient is found to have disease progression while on active therapy, the next blood draw will be on the first day of the next therapy and time point of subsequent blood draws will depend on the type of therapy the patient receives.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Whole blood will be collected using standard phlebotomy procedures

SUMMARY:
The primary objective of this study is to establish circulating tumor cell (CTC) derived xenografts and assess the activity of novel DNA repair inhibitors as a function of DNA repair mutations detected in CTC samples (personalize DNA repair therapy).

DETAILED DESCRIPTION:
There are 2 cohorts for this study. Cohort A & Cohort B are for patient subjects. Patients can participate in both cohorts simultaneously, or only one cohort per patient preference.

The investigators anticipate that most patients who participate in Cohort B will also participate in Cohort A because Cohort A only requires a one-time blood draw at baseline.

Cohort A: 20 patients with NSCLC and 20 patients with SCLC. Blood samples will be collected from eligible patients only once at baseline. These samples will be immediately processed for CTCs and CTC derived xenografts.

Cohort B: 15 patients with NSCLC and 15 patients with SCLC. Blood samples will be collected from eligible patients at baseline just prior to initiation of therapy. Samples will also be collected on day 1 of every cycle of therapy for 4 cycles (typical cycles are 21 days for chemotherapy, 28 days for targeted therapy and 14 days for immune therapy). At the time of initiation of the treatment break, blood samples will be collected. During the treatment break, patients will be followed every 6-12 weeks with imaging studies, and we will collect blood samples at each visit. At the time of disease progression in the event patient goes on best supportive care, the last blood draw will be at the time of this decision as there will unlikely be any further imaging studies going forward. If a patient is found to have disease progression while on active therapy, the next blood draw will be on the first day of the next therapy and time point of subsequent blood draws will depend on the type of therapy the patient receives. The goal is to define whether CTC loads whether CTC loads predict symptoms, response, and disease recurrence.

For Cohorts A & B: Investigators will make every attempt to time the blood collection to coincide with blood collection for therapeutic purposes in order to minimize discomfort. Blood sample collection will take place either in the outpatient clinic, or while inpatient (at IUSCCC, Indiana University Hospital, or Eskenazi hospital). Patients can participate in both cohorts simultaneously, or only one cohort per patient preference.

ELIGIBILITY:
Inclusion Criteria Cohort A (one-time blood sample) & Cohort B (multiple blood samples)

* Histologically or cytologically confirmed lung cancer (both non-small cell lung cancer and small cell lung cancer are allowed)
* Stage 4 NSCLC or extensive-stage SCLC
* Newly diagnosed disease with no prior systemic therapy for advanced disease Note: Patients that have received prior adjuvant chemotherapy or prior chemoradiotherapy for earlier stage lung cancer are allowed if treatment was completed ≥3 months.
* Age ≥ 18 years
* Ability to understand and the willingness to sign a written informed consent document

Inclusion of Women and Minorities Both men and women of all races and ethnic groups are eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll 2 cohorts for this study. Cohort A & Cohort B are for patient subjects. Patients can participate in both cohorts simultaneously, or only one cohort per patient preference. We anticipate that most patients who participate in Cohort B will also participate in Cohort A because Cohort A only requires a one-time blood draw at baseline.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-10-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Assess activity of novel DNA repair inhibitors as a function of DNA repair mutations detected in CTC samples | Baseline
  All analyses will be done by disease group (i.e., NSCLC and SCLC). For the primary objective, CTC derived xenografts will be generated, and CTCs will be analyzed for DNA repair defects, and used to evaluate the activity of novel DNA repair inhibitors. We will look at CTCs by group [specific DNA defect (yes or no), treated vs untreated] using histograms and compare groups statistically using two group Satterthwaite t-tests with a 0.050 two-sided significance level.

CONTACTS AND LOCATIONS:
Overall Officials: Shadia Jalal, MBBS, Principal Investigator — Indiana University School of Medicine, Indiana University Simon Cancer Center
Locations (2):
- United States (2):
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Roudebush VA Medical Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No